CLINICAL TRIAL: NCT05616104
Title: FLEX FIRST Registry Research Protocol
Status: Completed | Type: Observational
Sponsor: VentureMed Group Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VMG-2022-001
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Arteriovenous Fistula; Arteriovenous Graft; Fistula; Arterial Occlusive Diseases
MeSH Terms: conditions — Arteriovenous Fistula; Fistula; Arterial Occlusive Diseases | interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- FLEX Vessel Prep followed by angioplasty: Eligible subjects will be treated with the FLEX Vessel Prep system followed by balloon angioplasty.
  Interventions: Device: FLEX Vessel Prep System

INTERVENTIONS:
Device: FLEX Vessel Prep System — The FLEX Vessel Prep System to create circumferential, continuous micro-incisions along the length of the stenosis by performing a retrograde pullback through the lesion.
  Following FLEX, standard balloon angioplasty is performed with an uncoated PTA balloon sized to meet the reference vessel diameter, according to its corresponding Instructions for Use. Once advanced into the lesion, the balloon should be inflated according to the site's standard of care.
  Other Names: Balloon Angioplasty

SUMMARY:
Prospective, observational study evaluating the clinical use and outcomes of the FLEX Vessel Prep (VP) system in arteriovenous fistulae or grafts presenting with clinical or hemodynamic abnormalities following 12 months post treatment.

DETAILED DESCRIPTION:
Prospective, observational study evaluating the clinical use and outcomes of the FLEX Vessel Prep (VP) system in arteriovenous fistulae or grafts presenting with clinical or hemodynamic abnormalities in real-world subjects per the Institution's standard practice and at 1-, 6-, and 12-months following treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age.
2. Subject is currently scheduled to undergo an endovascular intervention of arteriovenous fistula or graft due to clinical and hemodynamic abnormalities meeting the KDOQI Guidelines for AV access dysfunction:

   * Elevated venous pressure during hemodialysis,
   * Abnormal physical findings, and
   * Unexplained decrease in delivered dialysis dose.
3. Subject has a reasonable expectation of remaining on hemodialysis for ≥12 months.
4. Subject is legally competent, informed of the study, voluntarily agrees to participate, and signs the informed consent form.
5. Subject understands the study and is willing and able to comply with the follow-up requirements.

Exclusion Criteria:

1. Subject has a known or suspected systemic infection.
2. Subject has a known or suspected infection of the hemodialysis graft.
3. Subject has an untreatable allergy to radiographic contrast material.
4. In the opinion of the operating physician, the subject's hemodialysis access is unsuitable for endovascular treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with AVF/AVG stenosis who are eligible for FLEX/Angioplasty treatment
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Target Lesion Primary Patency Rate | 6 months post procedure
  Defined as freedom from clinically driven target lesion re-intervention (CD-TLR) or access circuit thrombosis measured through 6-months post- procedure.
Serious Adverse Event Rate | 1 month
  Defined as the Serious Adverse Event (SAE) rate involving the AV access circuit through 1-month post-procedure.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Open Access Vascular Access, Miami, Florida
  - Minneapolis Vascular Surgery Center, New Brighton, Minnesota
  - Dialysis Access Institute, Orangeburg, South Carolina
  - Spartanburg Regional Health, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No